CLINICAL TRIAL: NCT06284733
Title: Whole-body Vibration Without Visual Feedback on Postural Steadiness in Unilateral Trans-femoral Traumatic Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, lectrurer of physical therapy for general surgery and dermatology, MTI University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004874
Record Dates: First submitted 2024-02-19; First posted 2024-02-29 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Amputation; Traumatic, Leg, Lower
Keywords: postural stability; amputee

STUDY DESIGN:
Intervention Model Description: They will be assigned into three equal groups:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (WBV group)(30 HZ,4 mm ,eyes open) (Experimental): This group includes 36 patients with unilateral trans-femoral traumatic amputation; they will receive WBV and conservative care.
  Interventions: Device: Whole-body vibration plus conservative care; Other: conservative care
- Group B (visual feedback-deprived and WBV (VFD WBV) (30 HZ,4 mm ,eyes close) (Experimental): This group includes 36 patients with unilateral trans-femoral traumatic amputation; they will receive visual feedback-deprived plus WBV (VFDWBV) and conservative care.
  Interventions: Device: Whole-body vibration plus conservative care; Other: conservative care
- Group C(control group (0 Hz, eyes open) (Sham Comparator): This group includes 36 patients with unilateral trans-femoral traumatic amputation; they will receive conservative care.
  Interventions: Other: conservative care

INTERVENTIONS:
Device: Whole-body vibration plus conservative care — Whole-body vibration (WBV) is a therapeutic method that exposes the entire body to mechanical oscillations while the patient stands or sits on a vibrating platform. This method was used in rehabilitation to improve muscle function, joint stability, balance control and to reduce the risk of falling.
  Arms: Group A (WBV group)(30 HZ,4 mm ,eyes open); Group B (visual feedback-deprived and WBV (VFD WBV) (30 HZ,4 mm ,eyes close)
Other: conservative care — 1. Stretching and ROM exercises daily to make sure that the patient can straighten hip; this makes walking, and even lying in bed, more comfortable.
  2. Resting hip on a pillow, as this promotes a hip flexion contracture
  3. A pillow between legs, as this lengthens the inner thigh muscle that helps to keep legs together while walking, and shortens the outer thigh muscles so that walking and standing with feet apart.
  4. Regular skin care.
  5. Regular prosthetic care.

SUMMARY:
This study will investigate the effects of Whole-body vibration without visual feedback on postural steadiness in unilateral trans-femoral traumatic amputees. This study will be carried out at the outpatient clinic of the faculty of physical therapy, modern university for technology and information, and El Wafaa wel Amal hospital.

All participants will sign a written consent form after receiving full information about the purpose of the study, procedure, possible benefits, privacy, and use of data.

DETAILED DESCRIPTION:
The postural steadiness is the dynamics of the postural control system associated with maintaining balance during quiet standing and usually assessed by the displacement of the centre of pressure (COP).

The control of posture is maintained by a complex sensory-motor system, which integrates information from the visual, proprioceptive, vestibular and somato-sensory systems. In the case of a unilateral trans femoral amputee, the individual becomes structurally asymmetrical, as there is an altered sensation and a loss of musculature on the amputated side. Whole-body vibration (WBV) is a therapeutic method that exposes the entire body to mechanical oscillations while the patient stands or sits on a vibrating platform. This method was used in rehabilitation to improve muscle function, joint stability, balance control and to reduce the risk of falling.

Whole-body vibration (WBV) training helps to improve the dysfunction of the nervous system and musculoskeletal system diseases, to prevent and relieve osteoporosis in the elderly, and to promote sports injury recovery and improve sports performance. But till now there is no judgment concerning the difference and significance of Whole-body vibration without visual feedback on postural steadiness in unilateral trans-femoral traumatic amputees.

ELIGIBILITY:
Inclusion Criteria:

* 40 to 55 years of age.
* Residual femoral length from ischial tuberosity to the end of the limb with distal soft tissue compressed (15-35 cm)
* Unilateral trans-femoral traumatic amputation with single-axis mechanical knees, axial foot (single axis).
* Able to walk without the use of any assistive device; subjects must have obtained a score of > 5 for Houghton Scale to indicate active use of prosthesis and > 41 for Berg Balance Scale (BBS).
* Medicare level 3 (community) ambulatory or above.
* Ability to descend stairs and hills without caregiver and assistive devices.
* Be able to independently provide informed consent.
* Be willing to comply with study procedures.

Exclusion Criteria:

* Reduced somatosensory sensibility of the non-affected limb, ulceration or pain at the stump
* the amputation was of vascular origin
* Poor fittings of prosthesis
* Visual or vestibular impairment (vertigo or dizziness)
* Lower limb musculoskeletal injury and other neurological deficits

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Prosthetic leg stability test | base line and after 12 weeks.
  Prior to testing, the subject will be asked to center the foot on the platform in a position that will be level and stable. This foot placement will maintained through -out all 3 trials for the prosthetic leg. This position will be used as the level reference point from which degree of displacement was measured. The subject will instructed to stand on foot with the knee slightly flexed (15°) on the platform, with the contralateral knee flexed to 90° for 20 seconds (test period). Level 8 will be selected for use during testing

SECONDARY OUTCOMES:
Sway Index | base line after 12 weeks
  The CTSIB (Modified Clinical Test of Sensory Interaction on Balance) is a standard test for postural steadiness on different surfaces. This test was designed to assess the patient's ability to integrate sensory information to maintain body equilibrium.
Limits of Stability Test | base line after 12 weeks
  The subjects will be asked to move directly toward the target, the best expected outcome was a straight path. During this test, 8 targets will be presented in each direction, and the subjects were randomly given instructions. The subjects will be requested to move their centre of gravity toward the targets, touch them, and then return to the center.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mohamed Ahmed Abdelhady, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elfeky HM, Elfahl AM, Mohamed HS. Whole-Body Vibration Without Visual Feedback on Postural Steadiness in Unilateral Trans-Femoral Traumatic Amputees: A Randomized Controlled Trial. Physiother Res Int. 2025 Apr;30(2):e70031. doi: 10.1002/pri.70031. PMID 39902775